CLINICAL TRIAL: NCT03225001
Title: Edwards SAPIEN XT Transcatheter Heart Valve Therapy for Patients With a Failing Aortic Bioprosthetic Valve
Brief Title: PARTNER II Trial: Placement of AoRTic TraNscathetER Valves II - Nested Registry 3/Valve-in-Valve
Acronym: PII NR3/ViV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-12 NR3/ViV
Record Dates: First submitted 2017-07-17; First posted 2017-07-21 (Actual); Results first posted 2018-01-09 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-02

CONDITIONS: Aortic Stenosis; Cardiomyopathy, Hypertrophic
Keywords: SAPIEN XT; Partner II; cardiovascular disease; heart disease; aortic disease; SAVR; TAVR; failing surgical valve; failing valve; failing bioprosthetic valve
MeSH Terms: conditions — Aortic Valve Stenosis; Cardiomyopathy, Hypertrophic; Cardiovascular Diseases; Heart Diseases; Aortic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Failing surgical valve (Experimental): Patients with a failing surgical bioprosthetic valve in the aortic position demonstrating stenosis and/or insufficiency will be treated with Edwards SAPIEN XT transcatheter valve.
  Interventions: Device: Edwards SAPIEN XT transcatheter valve, Model 9300TFX

INTERVENTIONS:
Device: Edwards SAPIEN XT transcatheter valve, Model 9300TFX — Edwards SAPIEN XT THV system Model 9300TFX with the associated delivery systems.
  Other Names: TAVI

SUMMARY:
To assess the safety and effectiveness of the SAPIEN XT transcatheter heart valve in patients with a failing surgical aortic bioprosthetic valve.

DETAILED DESCRIPTION:
A prospective, single-arm, multicenter clinical trial. The trial will enroll patients with a failing surgical bioprosthetic valve in the aortic position demonstrating stenosis and/or insufficiency. This is a PARTNER II nested registry.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has senile degenerative aortic valve stenosis with echocardiographically derived criteria: mean gradient >40 mmHg or jet velocity greater than 4.0 m/s and an initial aortic valve area (AVA) of ≤0.8 cm2 or indexed EOA < 0.5 cm2/m2. Qualifying echo must be within 60 days of the date of the procedure.
2. Patient was symptomatic from his/her aortic valve stenosis, as demonstrated by NYHA Functional Class II or greater.
3. The heart team agreed (and verified in the case review process) that valve implantation would likely benefit the patient.
4. The study patient or the study patient's legal representative was informed of the nature of the study, agreed to its provisions and had provided written informed consent as approved by the Institutional Review Board (IRB) of the respective clinical site.
5. Heart team consensus that the risk of surgical mortality or major morbidity ≥ 50%.
6. Stenosed or insufficient surgically implanted bioprosthetic valve in the aortic position.

Exclusion Criteria:

1. Bioprosthetic valve labeled external diameter < 21mm.
2. Surgical or transcatheter valve in another position on the same side of the heart (mitral and tricuspid rings are not an exclusion).
3. Infectious endocarditis within 6 months.
4. Acute myocardial infarction ≤ 1 month (30 days) before the intended treatment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2012-06-11 (Actual); Primary Completion 2016-12-16 (Actual); Study Completion 2020-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Webb, MD, Principal Investigator — St. Paul's Hospital, Vancouver, British columbia, Canada; Michael Mack, MD, Principal Investigator — Baylor Heart Hospital, Plano, TX
Locations (47):
- United States (46):
  - Scripps Green Hospital, La Jolla, California
  - Scripps Memorial Hospital, La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Mercy General Hospital, Sacramento, California
  - Stanford University Medical Center, Stanford, California
  - University of Colorado Hospital, Denver, Colorado
  - Washington Hospital Center (WHC), Washington D.C., District of Columbia
  - Morton Plant Hospital, Clearwater, Florida
  - University of Miami, Miami, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Northwestern Hospital, Chicago, Illinois
  - NorthShore University HealthSystem Research Institute, Evanston, Illinois
  - Prairie Education and Research Cooperative, Springfield, Illinois
  - The University of Iowa, Iowa City, Iowa
  - University of Louisville Jewish Hospital, Louisville, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Mayo Clinic-Saint Marys Hospital, Rochester, Minnesota
  - Saint Luke's Hospital of Kansas City Mid America, Kansas City, Missouri
  - Washington University - Barnes Jewish Hospital, St Louis, Missouri
  - Nebraska Heart Institute, Lincoln, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Winthrop-University Hospital, Mineola, New York
  - Cornell University, New York, New York
  - Columbia University Medical Center/ New York Presbyterian Hospital, New York, New York
  - East Carolina Heart Institute at East Carolina University, Greenville, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - Providence St.Vincent Medical Center, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - The Heart Hospital Baylor Plano, Dallas, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - The University of Texas Health Science Center at Houston/Memorial Hermann Texas Medical Center, Houston, Texas
  - Intermountain Medical Center, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - University of Washington, Seattle, Washington
  - University of Wisconsin - Madison, Madison, Wisconsin
- St. Paul's Hospital, Providence Health Care, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shahim B, Redfors B, Lindman BR, Chen S, Dahlen T, Nazif T, Kapadia S, Gertz ZM, Crowley AC, Li D, Thourani VH, Kodali SK, Zajarias A, Babaliaros VC, Guyton RA, Elmariah S, Herrmann HC, Cohen DJ, Mack MJ, Smith CR, Leon MB, George I. Neutrophil-to-Lymphocyte Ratios in Patients Undergoing Aortic Valve Replacement: The PARTNER Trials and Registries. J Am Heart Assoc. 2022 Jun 7;11(11):e024091. doi: 10.1161/JAHA.121.024091. Epub 2022 Jun 3. PMID 35656983
- [Derived] Webb JG, Murdoch DJ, Alu MC, Cheung A, Crowley A, Dvir D, Herrmann HC, Kodali SK, Leipsic J, Miller DC, Pibarot P, Suri RM, Wood D, Leon MB, Mack MJ. 3-Year Outcomes After Valve-in-Valve Transcatheter Aortic Valve Replacement for Degenerated Bioprostheses: The PARTNER 2 Registry. J Am Coll Cardiol. 2019 Jun 4;73(21):2647-2655. doi: 10.1016/j.jacc.2019.03.483. PMID 31146808

RESULTS

PARTICIPANT FLOW:
Groups:
- Edwards SAPIEN XT THV in Patients With Failing SAVR: Patients with a failing surgical bioprosthetic valve (SAVR) in the aortic position demonstrating stenosis and/or insufficiency will be treated with Edwards SAPIEN XT transcatheter valve.
  Edwards SAPIEN XT transcatheter valve, Model 9300TFX: Edwards SAPIEN XT THV system Model 9300TFX with the associated delivery systems.
Period: Overall Study
Arm/Group | Edwards SAPIEN XT THV in Patients With Failing SAVR
Started | 197
Valve-Implanted | 195
Completed | 188
Not Completed | 9

BASELINE CHARACTERISTICS:
Arm/Group | Edwards SAPIEN XT THV in Patients With Failing SAVR
Number analyzed (Participants) | 197
Age, Continuous [Mean (Standard Deviation); unit: Years] | 78.5 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78
  Male | 119
STS Score [Mean (Standard Deviation); unit: units on a scale] — The Society of Thoracic Surgeons (STS) score measures patient risk at the time of cardiovascular surgery on a scale that ranges from 0% to 100%, with higher numbers indicating greater risk.
  units on a scale | 9.7 (5.1)
NYHA III/IV [Count of Participants; unit: Participants] — New York Heart Association (NYHA), functional classification of heart failure based on how much a patient is limited during physical activity. The rating ranges from I - IV, with the lowest as no limitations and the highest unable to carry on any physical activity without discomfort.
  Participants | 188

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With All-Cause Mortality, All Stroke, Moderate or Severe Obstruction, or Moderate or Severe Paravalvular Leak (Composite)
Description: The primary endpoint of all-cause mortality, all stroke, moderate or severe obstruction, or moderate or severe paravalvular leak
Time Frame: 30-day
Population: Twenty-nine patients had missing echocardiography data.
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards SAPIEN XT THV in Patients With Failing SAVR
Number analyzed (Participants) | 166
Participants | 28

2. Secondary Outcome: Number of Participants With Mortality From Any Cause
Description: Cardiovascular cause is also included
Time Frame: 30 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards SAPIEN XT THV in Patients With Failing SAVR
Number analyzed (Participants) | 195
Participants | 8

ADVERSE EVENTS:
Time Frame: 30-day
Description: Site reported events Only Valve-Implant patients are analyzed.
Arm/Group | Edwards SAPIEN XT THV in Patients With Failing SAVR
All-Cause Mortality (participants affected / at risk) | 8/195
Serious Adverse Events (participants affected / at risk) | 109/195
Other Adverse Events (participants affected / at risk) | 142/195
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Edwards SAPIEN XT THV in Patients With Failing SAVR (N=195)
Abnormal Lab Value (Investigations) | 3 (3)
Anemia/Hemolytic Anemia (Vascular disorders) | 3 (4)
Angina/Cardiac Chest Pain (Cardiac disorders) | 4 (5)
Arrhythmia/Conduction System Injury (Defect) (Cardiac disorders) | 11 (12)
Bacteremia (Infections and infestations) | 6 (8)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4)
Cardiac Arrest (Cardiac disorders) | 5 (5)
Cardiogenic Shock (Cardiac disorders) | 1 (1)
Change in level of consciousness (Nervous system disorders) | 1 (1)
Compartment syndrome (Injury, poisoning and procedural complications) | 1 (1)
Coronary Flow Obstruction/Transvalvular flow disturbance (Injury, poisoning and procedural complications) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (7)
Embolization including air/calcific valve material or Thrombus (Injury, poisoning and procedural complications) | 1 (1)
Encephalopathy (Nervous system disorders) | 2 (2)
Endocarditis (Infections and infestations) | 1 (1)
Failure of percutaneous access site closure resulting in intervention (Injury, poisoning and procedural complications) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 6 (6)
Gastro Intestinal Event (Gastrointestinal disorders) | 5 (6)
Gastro Intestinal Event Nonhemorrhagic (Gastrointestinal disorders) | 6 (7)
Genito Urinary Event (Renal and urinary disorders) | 1 (1)
Genito Urinary Event Nonhemorrhagic (Renal and urinary disorders) | 1 (1)
Heart Failure / CHF / Low output Failure (Cardiac disorders) | 26 (28)
Hemorrhage (Vascular disorders) | 22 (22)
Hemorrhagic Stroke (Nervous system disorders) | 2 (2)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 3 (3)
Ischemic Stroke (Vascular disorders) | 4 (5)
Mitral Valve Injury or Insufficiency (Injury, poisoning and procedural complications) | 1 (1)
Multi Organ Failure (Investigations) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 3 (3)
Non Structural Dysfunction (Injury, poisoning and procedural complications) | 3 (3)
Pain (Nervous system disorders) | 7 (7)
Perforation (Injury, poisoning and procedural complications) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pseudoaneurysm (Vascular disorders) | 1 (1)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pulmonary Effusion (Respiratory, thoracic and mediastinal disorders) | 9 (10)
Renal Failure (Renal and urinary disorders) | 9 (10)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 18 (19)
Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Restenosis (Vascular disorders) | 3 (3)
Rupture (Injury, poisoning and procedural complications) | 1 (1)
Sepsis (Infections and infestations) | 8 (8)
Syncope (Vascular disorders) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Unknown cause of Death (Investigations) | 4 (4)
Other (Investigations) | 15 (18)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Undetermined Stroke (Investigations) | 1 (1)
TIA (Vascular disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (4)
Confusion (Psychiatric disorders) | 2 (2)
Access site infection (Infections and infestations) | 1 (1)
Cough (Infections and infestations) | 1 (1)
Dementia (Psychiatric disorders) | 1 (2)
Device Migration/malposition requiring intervention (Injury, poisoning and procedural complications) | 2 (2)
Drug Reaction (Investigations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Edwards SAPIEN XT THV in Patients With Failing SAVR (N=195)
Abnormal Lab Value (Investigations) | 23 (39)
Anemia/Hemolytic Anemia (Injury, poisoning and procedural complications) | 23 (24)
Arrhythmia/Conduction System Injury (Defect) (Cardiac disorders) | 38 (42)
Fall (Injury, poisoning and procedural complications) | 12 (13)
Heart Failure / CHF / Low output Failure (Cardiac disorders) | 12 (12)
Hemorrhage (Vascular disorders) | 40 (45)
Hypotension (Vascular disorders) | 10 (10)
Pain (Nervous system disorders) | 12 (19)
Pulmonary Effusion (Respiratory, thoracic and mediastinal disorders) | 11 (12)
Renal Insufficiency or Renal Failure (Renal and urinary disorders) | 16 (20)
Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 16 (16)
Thrombocytopenia (Blood and lymphatic system disorders) | 23 (23)
Urinary Tract Infection (Infections and infestations) | 18 (18)
Other (Investigations) | 50 (63)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No